Title: "Assessing the Efficacy of IV Ibuprofen for Treatment of Pain in Orthopedic Trauma Patients."

NCT02152163

**Document Date: September 6, 2019** 

## **Statistical Analysis**

The primary efficacy endpoint regarding the amount of opioid medication was analyzed using the difference in least squares means (LS Means) from an analysis of covariance (ANCOVA) model with a fixed effect for treatment and baseline pain intensity as a covariate. PID was analyzed using the same ANCOVA model. The secondary efficacy endpoints of length of hospital stay and time to first narcotic medication were analyzed using the Kaplan-Meier estimation method. A Cox proportional hazards regression analysis with effects for treatment and baseline pain intensity was performed to determine the hazard ratio (HR), the corresponding 95% CI, and to compare the treatment groups. For the comparison of baseline tobacco, alcohol, recreational drugs and pain medication usage between groups,  $\chi 2$  analysis was used with p <0.05 considered as statistically significantly different. Treatment assignment (Placebo or Caldolor®) remained blind to all authors, until all results were obtained, and all statistical analysis had been completed.